CLINICAL TRIAL: NCT04708782
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of the Efficacy and Safety of Inhaled Treprostinil in Subjects With Idiopathic Pulmonary Fibrosis (TETON-1)
Brief Title: Study of Efficacy and Safety of Inhaled Treprostinil in Subjects With Idiopathic Pulmonary Fibrosis
Acronym: TETON-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN-PF-301
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease
Keywords: Treprostinil; IPF; ILD
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo inhaled using an ultrasonic nebulizer QID
  Interventions: Drug: Placebo; Device: Treprostinil Ultrasonic Nebulizer
- Inhaled Treprostinil (Experimental): Treprostinil for inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath. Inhaled QID and titrated up to a target of 12 breaths QID or until the subject reaches their maximum clinically tolerated dose.
  Interventions: Drug: Inhaled Treprostinil; Device: Treprostinil Ultrasonic Nebulizer

INTERVENTIONS:
Drug: Placebo — Placebo administered QID
  Arms: Placebo
Drug: Inhaled Treprostinil — Inhaled treprostinil (6 mcg/breath) administered QID
  Other Names: Tyvaso
  Arms: Inhaled Treprostinil
Device: Treprostinil Ultrasonic Nebulizer — Treprostinil ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath.

SUMMARY:
Study RIN-PF-301 is designed to evaluate the superiority of inhaled treprostinil against placebo for the change in absolute forced vital capacity (FVC) from baseline to Week 52.

DETAILED DESCRIPTION:
Study RIN-PF-301 is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the superiority of inhaled treprostinil against placebo for the change in absolute FVC in subjects with IPF over a 52-week period. Subjects will be randomly allocated 1:1 to receive inhaled treprostinil or placebo. All subjects will initiate inhaled treprostinil or placebo at a dose of 3 breaths administered 4 times daily (QID) and will titrate to a target dosing regimen of 12 breaths QID. Study drug doses may be titrated up as tolerated, until the target dose or maximum clinically tolerated dose is achieved. Once eligible, 6 Treatment Period visits to the clinic will be required at Weeks 4, 8, 16, 28, 40, and 52.

Efficacy assessments include spirometry (FVC), time to clinical worsening, time to first acute exacerbation of IPF, overall survival, King's Brief Interstitial Lung Disease (K-BILD) questionnaire, plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) concentration, supplemental oxygen use, and lung diffusion capacity (DLCO). Safety assessments include the development of adverse events (AEs)/serious adverse events (SAEs), vital signs, clinical laboratory parameters, and electrocardiogram (ECG) parameters.

Subjects who complete the Week 52 Visit may be offered the opportunity to enter an open-label extension (OLE) study after completing the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject gives voluntary informed consent to participate in the study.
2. Subject is ≥40 years of age, inclusive, at the time of signing informed consent.
3. The subject has a diagnosis of IPF based on the 2018 ATS/ERS/JRS/ALAT Clinical Practice Guideline (Raghu 2018) and confirmed by central review of high-resolution computed tomography (HRCT) (performed within the previous 12 months), and if available, surgical lung biopsy.
4. FVC ≥45% predicted at Screening.
5. Subjects on pirfenidone or nintedanib must be on a stable and optimized dose for ≥30 days prior to Baseline. Concomitant use of both pirfenidone and nintedanib is not permitted.
6. Women of childbearing potential must be non-pregnant (as confirmed by a urine pregnancy test at Screening and Baseline) and non-lactating, and will abstain from intercourse (when it is in line with their preferred and usual lifestyle) or use 2 medically acceptable, highly effective forms of contraception for the duration of the study, and at least 30 days after discontinuing study drug.
7. Males with a partner of childbearing potential must use a condom for the duration of treatment and for at least 48 hours after discontinuing study drug.
8. In the opinion of the Investigator, the subject is able to communicate effectively with study personnel, and is considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

1. Subject is pregnant or lactating.
2. Subject has primary obstructive airway physiology: FEV1/FVC <0.70 at Screening.
3. The subject has shown intolerance or significant lack of efficacy to a prostacyclin or prostacyclin analogue that resulted in discontinuation or inability to effectively titrate that therapy.
4. The subject has received any PAH-approved therapy, including prostacyclin therapy (epoprostenol, treprostinil, iloprost, or beraprost; except for acute vasoreactivity testing), IP receptor agonists (selexipag), endothelin receptor antagonists, phosphodiesterase type 5 inhibitors (PDE5-Is), or soluble guanylate cyclase stimulators within 60 days prior to Baseline. As needed use of a PDE5-I for erectile dysfunction is permitted, provided no doses are taken within 48 hours of any study-related efficacy assessments.
5. Use of any of the following medications: azathioprine (AZA), cyclosporine, mycophenolate mofetil, tacrolimus, oral corticosteroids (OCS) >20 mg/day or the combination of OCS+AZA+N-acetylcysteine within 30 days prior to Baseline; cyclophosphamide within 60 days prior to Baseline; or rituximab within 6 months prior to Baseline.
6. The subject is receiving >10 L/min of oxygen supplementation by any mode of delivery at rest at Baseline.
7. Exacerbation of IPF or active pulmonary or upper respiratory infection within 30 days prior to Baseline. Subjects must have completed any antibiotic or steroid regimens for treatment of the infection or acute exacerbation more than 30 days prior to Baseline to be eligible. If hospitalized for an acute exacerbation of IPF or a pulmonary or upper respiratory infection, subjects must have been discharged more than 90 days prior to Baseline to be eligible.
8. Uncontrolled cardiac disease, defined as myocardial infarction within 6 months prior to Baseline or unstable angina within 30 days prior to Baseline.
9. In the opinion of the Investigator, the subject has any condition that would interfere with the interpretation of study assessments or would impair study participation or cooperation.
10. Use of any other investigational drug/device or participation in any investigational study in which the subject received a medical intervention (ie, procedure, device, medication/supplement) within 30 days prior to Screening. Subjects participating in non-interventional, observational, or registry studies are eligible.
11. Life expectancy <6 months due to IPF or a concomitant illness.
12. Acute pulmonary embolism within 90 days prior to Baseline.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Change in Absolute FVC from Baseline to Week 52 | Baseline to Week 52
  The FVC measurement indicates the amount of air a person can forcefully and quickly exhale after taking a deep breath.

SECONDARY OUTCOMES:
Time to Clinical Worsening | Baseline to Week 52
  Clinical worsening was monitored from randomization until 1 of the following criteria were met: death (all causes), hospitalization due to a respiratory indication, or 10% relative decline in % predicted FVC.
Time to First Acute Exacerbation of IPF | Baseline to Week 52
  An exacerbation of IPF is defined as an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality.
Overall Survival at Week 52 | Week 52
  Vital status will be assessed for all subjects at Week 52, including those who discontinue the study prematurely or who withdraw consent.
Change in % Predicted FVC from Baseline to Week 52 | Baseline to Week 52
  The FVC measurement indicates the amount of air a person can forcefully and quickly exhale after taking a deep breath. Percent predicted FVC is calculated based on factors such as ethnicity, sex, age, height, and weight.
Change in K-BILD Questionnaire Score from Baseline to Week 52 | Baseline to Week 52
  The K-BILD is a self-administered, 15-item questionnaire validated for patients with interstitial lung disease (ILD) consisting of 3 domains (breathlessness and activities, psychological, and chest symptoms).
Change in DLCO from Baseline to Week 52 | Baseline to Week 52
  The DLCO measurement measures how well oxygen moves from the lungs to the blood.

CONTACTS AND LOCATIONS:
Locations (99):
- United States (91):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center-Phoenix, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center - Norton Thoracic Institute, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - UC San Diego Health, La Jolla, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - NewportNativeMD, Inc, Newport Beach, California
  - University of California, Irvine, Orange, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - UC Davis Health Medical Center, Sacramento, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - St. Francis Sleep Allergy & Lung Institute, Clearwater, Florida
  - University of Florida Health at Shands, Gainesville, Florida
  - Ascension St. Vincent's, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Pulmonary Disease Specialists, PA d/b/a PDS Research, Kissimmee, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Coastal Pulmonary & Critical Care PLC, St. Petersburg, Florida
  - University of South Florida Health, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Healthcare Atlanta, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center Outpatient Pulmonary Clinic, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Community Health Network, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - LSU Health Sciences Center New Orleans, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - LSU Health Science Center Shreveport, Shreveport, Louisiana
  - Johns Hopkins Asthma & Allergy Center, Baltimore, Maryland
  - Adventist Healthcare White Oak Medical CEnter, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Int Med Pulmonary and critical care, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Lung Research Center, Chesterfield, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Creighton University Clinical Research Office, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - St Joseph's Physician's Pulmonary Health, Liverpool, New York
  - Northwell Health, New Hyde Park, New York
  - University of Rochester Medical center, Rochester, New York
  - Stony Brook Advanced Specialty Care, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - PulmonIx, LLC, Greensboro, North Carolina
  - East Carolina University and Leo Jenkins Cancer Center, Greenville, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - Martha Morehouse Medical Pavilion, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Oregon Clinic, PC, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center/Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thoams Jefferson,Hospital University, Philadelphia, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Midlands, Columbia, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Statecare Pulmonary Consultants, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Univrsity of Texas Southwestern Medical Center, Dallas, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - Baylor Clinic-Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - A & A Research Consultants, LLC, McAllen, Texas
  - Metroplex Pulmonary and Sleep Center PA, McKinney, Texas
  - Renovatio Clinical Consultants, LLC, The Woodlands, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - University of Wisconsin School of Medicine and Public health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - St.Paul's Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement Limited, Ajax, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec-Universite, Québec, Quebec
  - Centre d'investigation Clinique Mauricie, Trois-Rivières, Quebec
- Chile (2):
  - Centro Respiratorio Integral LTDA. (CENRESIN), Quillota, Región de Valparaíso
  - Fundacion Medica San Cristobal, Santiago, Santiago Metropolitan